CLINICAL TRIAL: NCT07379307
Title: THE EFFECT OF DİFFERENT MATERNAL POSİTİONS APPLİED DURİNG FETAL MONİTORİNG ON PAİN AND COMFORT LEVELS İN OBESE PREGNANT WOMEN
Brief Title: EFFECT OF DİFFERENT POSİTİONS ON PAİN AND COMFORT DURİNG FETAL MONİTORİNG İN OBESE PREGNANT WOMEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, hatice melike, Master's Student, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TUBITAK-2209A-1919B012309536; TUBITAK 2209-A (Other: The Scientific and Technological Research Council of Turkey (TUBITAK))
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Obesity in Pregnancy; Maternal Comfort During Fetal Monitoring
Keywords: electronic fetal monitoring; maternal obesity; comfort; pain
MeSH Terms: conditions — Pregnancy in Obesity; Pain | interventions — Supine Position; Palliative Care

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of three parallel groups. Each participant underwent fetal monitoring in a single maternal position. Pain and comfort levels were assessed during the monitoring procedure, and outcomes were compared between groups.
Masking Description: This is an open-label study. No participants, investigators, or outcome assessors were masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supported Left Lateral Position (Experimental): Participants underwent electronic fetal monitoring while lying in a supported left lateral position using pillows for positioning support.
  Interventions: Behavioral: Maternal Positioning during NST
- Unsupported Left Lateral Position (Experimental): Participants underwent electronic fetal monitoring while lying in an unsupported left lateral position without additional positioning aids.
  Interventions: Behavioral: Maternal Positioning during NST
- Supine Position (Experimental): Participants underwent electronic fetal monitoring while lying in the supine (back-lying) position.
  Interventions: Behavioral: Maternal Positioning during NST

INTERVENTIONS:
Behavioral: Maternal Positioning during NST — This intervention involves placing pregnant women at 28-40 weeks of gestation in specific positions (supported left lateral, supine, or left lateral without support) during Non-Stress Test (NST) monitoring. Each participant remains in the assigned position for 20-40 minutes while fetal heart rate is recorded using EFM. Pain/discomfort and overall comfort are assessed using Visual Analog Scale (VAS) and General Comfort Scale immediately after the intervention. The intervention is distinguished from other studies by the randomized allocation of three positional groups and simultaneous evaluation of maternal comfort and fetal monitoring outcomes.
  Other Names: Supported Left Lateral Position (Group 1); Supine Position (Group 2); Left Lateral without Support (Group 3)

SUMMARY:
This study was conducted to understand how different body positions during fetal monitoring affect pain and comfort in obese pregnant women. Fetal monitoring is a routine procedure used during pregnancy to check the baby's well-being. During this procedure, pregnant women are usually asked to lie still for a period of time, which may cause discomfort, especially for women with obesity.

The study included obese pregnant women in their third trimester who attended obstetrics outpatient clinics and underwent routine fetal monitoring. During the monitoring process, women were placed in one of three different positions: supported left side-lying, unsupported left side-lying, or lying on the back. Pain and comfort levels were assessed during and immediately after the fetal monitoring procedure.

The aim of this study was to determine which position provides greater comfort and less pain for obese pregnant women during fetal monitoring. The findings of this study may help health care professionals choose more comfortable positioning options and improve the overall pregnancy care experience for obese pregnant women.

DETAILED DESCRIPTION:
Fetal monitoring is a commonly used procedure during pregnancy to assess fetal well-being by recording the fetal heart rate and uterine activity. Although it is a routine and non-invasive procedure, remaining in the same position for an extended period of time may cause discomfort and pain, particularly in obese pregnant women. Maternal obesity is known to increase physical strain and may negatively affect comfort during clinical procedures.

This study was designed to evaluate the effects of different maternal positions applied during fetal monitoring on pain and comfort levels in obese pregnant women. The study was conducted with pregnant women who met the inclusion criteria and attended obstetrics outpatient clinics for routine fetal monitoring. Participants were assigned to one of three maternal positions during the monitoring process: supported left side-lying, unsupported left side-lying, or supine position.

During the fetal monitoring procedure, participants' pain and comfort levels were assessed using appropriate measurement methods. The primary focus of the study was to compare maternal comfort and pain perception across different positions during fetal monitoring. Understanding how positioning affects maternal comfort may contribute to improved clinical practices and enhance the quality of care provided to obese pregnant women during routine prenatal monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who voluntarily agree to participate in the study
* Aged between 19 and 40 years
* Experiencing a healthy pregnancy
* Gestational age between 28+0 and 40+0 weeks (only third-trimester pregnancies are included, as EFM monitoring is recommended after 27 weeks)
* Singleton pregnancy with a live fetus
* Body Mass Index (BMI) of 30 or higher
* No physical disabilities
* Able to speak Turkish to answer questions accurately
* No cognitive, comprehension, or communication difficulties

Exclusion Criteria:

* Pregnant women who do not agree to participate in the study
* Aged under 19 years or 41 years and above (adolescent and advanced-age pregnancies are excluded due to increased risk)
* Diagnosed with high-risk pregnancy
* Illiterate or unable to read/write
* Having a contagious disease
* Having a mental disorder or history of a mental disorder requiring treatment
* Having physical disabilities affecting mobility, hearing, or psychological function
* Gestational age less than 28+0 weeks
* Currently in active labor

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Maternal Comfort during NST | Immediately after NST
  Maternal overall comfort during Non-Stress Test (NST) will be assessed using the General Comfort Scale (Short Form). The scale consists of 28 items evaluating three sub-dimensions: relief, ease, and transcendence. Each item is rated on a 6-point Likert scale, where 1 indicates low comfort and 6 indicates high comfort. The assessment will be conducted immediately after the NST while the participant remains in the assigned position (supported left lateral, supine, or left lateral without support). This measure evaluates the effect of maternal positioning on overall comfort during fetal monitoring."

SECONDARY OUTCOMES:
General Comfort Scale Score | Immediately after NST
  Maternal overall comfort during Non-Stress Test (NST) will be assessed using the General Comfort Scale (Short Form). The scale consists of 28 items evaluating three sub-dimensions: relief, ease, and transcendence. Each item is rated on a 6-point Likert scale, where 1 indicates low comfort and 6 indicates high comfort. The assessment will be conducted immediately after the NST while the participant remains in the assigned position (supported left lateral, supine, or left lateral without support). This measure evaluates the effect of maternal positioning on overall comfort during fetal monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: demet çakır, Assistant Professor, Principal Investigator — Tokat Gaziosmanpaşa University, Department of Midwifery; Hatice melike evrin, Master's Student, Principal Investigator — Tokat Gaziosmanpaşa University, Department of Midwifery
Locations (1):
- Tokat State Hospital, Department of Obstetrics and Gynecology, NST Room, Tokat Province, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data from the Visual Analog Scale (VAS) and General Comfort Scale assessments will be shared, including participant age, gestational week, and body mass index (BMI). Data will be de-identified to protect participant privacy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified IPD and supporting information will be available from March 1, 2026, for a period of 2 years, upon reasonable request.
Access Criteria: De-identified individual participant data (VAS scores, General Comfort Scale results, age, gestational week, BMI) along with study protocol, informed consent form, and data dictionary/codebook will be available to other researchers upon reasonable request. Access will be granted after approval by the study principal investigator via secure data sharing platform or email.

REFERENCES:
- [Result] Evrin HM, Demet B; Effects of Maternal Position on Fetal Comfort during NST; Presented at the 2023 Kocaeli Midwifery Congress, Turkey; Unpublished
- See also: Related Info — https://example.com